CLINICAL TRIAL: NCT00860951
Title: P300 Brain Computer Interface Keyboard to Operate Assistive Technology
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jane Huggins, PhD, Research Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H0002 - AT P300 Keyboard Study; 5R21HD054697 (NIH); H133G090005 (Other Grant/Funding Number: Department of Education)
Record Dates: First submitted 2009-03-11; First posted 2009-03-13 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-05

CONDITIONS: Healthy; Amyotrophic Lateral Sclerosis; Neuromuscular Disease; Spinal Cord Injury; Cerebral Palsy
Keywords: Normal
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuromuscular Diseases; Spinal Cord Injuries; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brain Computer Interface Keyboard (Other): What effect does the environment (BCI, AT device, Computer) have on the accuracy of typing using a BCI keyboard?
  Interventions: Device: Brain Computer Interface Keyboard

INTERVENTIONS:
Device: Brain Computer Interface Keyboard — Subjects will wear an EEG cap for 1-4 hours (1-2 hours typical) per session and use the brain-computer interface to operate assistive technology. Subjects will be asked to participate in 3 sessions.

SUMMARY:
The purpose of this research is to develop tools enable people who are paralyzed to operate technology and access computers. These tools are called brain computer interfaces (BCIs). BCIs would let a person use brain signals to operate technology.

DETAILED DESCRIPTION:
The purpose of this research is to develop tools to help people who are paralyzed. These tools are called brain computer interfaces (BCIs). BCIs would let a person use brain signals to operate technology. The investigators want to make a BCI that can be used to operate commercially available technologies for communication, environmental control or computer access. The BCI would replace a keyboard to let people operate these technologies without moving. However, the investigators need people to test the BCI so that the investigators can see how well it can replace a keyboard. The investigators want to understand how well it can work so that the investigators can make it useful for people who are paralyzed. The investigators will ask people to use the BCI to do things like make a communication system speak or type words on a computer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Able to read text on a computer screen
* Able to understand and remember instructions concerning participation

Exclusion Criteria:

* Unable give informed consent.
* Unable to understand and follow instructions.
* Have abnormal tone or uncontrolled movements in the head-and-neck that would interfere with EEG recordings.
* Known to have photosensitive epilepsy.
* Open head lesions or sores

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Huggins, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan Direct Brain Interface Project, Ann Arbor, Michigan
  - Wadsworth Center, Albany, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brain Computer Interface Keyboard
Started | 29
Completed | 22
Not Completed | 7
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol.
Arm/Group | Brain Computer Interface Keyboard
Number analyzed (Participants) | 22
Age, Continuous [Mean (Full Range); unit: years] | 43 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Typing With BCI Keyboard.
Description: Accuracy for the sentence typed in each environment was calculated as the percentage of characters for which the result character matched the target character. The target characters were determined based on the next character needed to complete the sentence to be copied. In the case of errors, the next character was therefore a backspace to correct the error. The target characters were modified by subject comments to account for errors in selecting the next character.
  Once sentence was typed in each environment in each session on a separate day. From the three repeated sessions, there were therefore 9 total sentences per subject with 3 measures for each environment. These were treated as repeated measures for the analysis.
Time Frame: mean score from 3 sessions over 29 days
Measure: Mean (Full Range); unit: percentage accuracy
Groups:
- BCI Environment: Average accuracy of selections for three sessions of text copying within the BCI as a stand-alone device.
- Computer Environment: Average accuracy of selections for three sessions of text copying within the BCI acting as a keyboard replacement for a laptop computer.
- Assistive Technology Enironment: Average accuracy of selections for three sessions of text copying with the BCI acting as a keyboard replacement for a communication system.
Arm/Group | BCI Environment | Computer Environment | Assistive Technology Enironment
Number analyzed (Participants) | 22 | 22 | 22
percentage accuracy | 85 [35 to 100] | 83 [27 to 100] | 83 [36 to 100]

ADVERSE EVENTS:
Arm/Group | Brain Computer Interface Keyboard
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No